CLINICAL TRIAL: NCT05058339
Title: Distress Associated with Coronavirus Disease 2019 and Telehealth on Supportive Care Patients with Advanced Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1196; NCI-2021-09080 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1196 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-14; First posted 2021-09-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Advanced Malignant Solid Neoplasm; COVID-19 Infection; Hematopoietic and Lymphoid Cell Neoplasm; Locally Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm; Recurrent Hematologic Malignancy; Recurrent Malignant Solid Neoplasm
MeSH Terms: conditions — COVID-19; Hematologic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (survey): Patients complete survey over 20 minutes.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Complete survey

SUMMARY:
This study assesses the level of distress felt by cancer patients due to the coronavirus disease 2019 (COVID-19) pandemic. Researchers also want to learn if patients prefer to receive supportive care (palliative care) in person or through telemedicine (visits by phone or video call, such as Zoom). Information from this study may help doctors better understand how COVID-19 has affected patients with advanced cancer, patients' perceptions of telehealth, and may help clinicians tailor care to patients' needs during the pandemic.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess advanced cancer patients' level of distress due to the COVID-19 pandemic.

II. Assess patients' overall preference towards palliative telemedicine vs in person visits during the COVID-19 pandemic.

SECONDARY OBJECTIVES:

I. Assess associations between patient characteristics and perceptions of overall distress due to the COVID-19 pandemic.

II. Assess associations between patient characteristics and their attitudes and beliefs towards palliative telemedicine during the COVID-19 pandemic.

III. Compare the attitudes and beliefs towards palliative telemedicine between patients who completed visits via video vs telephone.

OUTLINE:

Patients complete survey over 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced cancer, defined as locally advanced, recurrent or metastatic disease
* Age 18 or greater
* Patient presenting for at least two follow-up visits with Supportive Care visit since the COVID19 pandemic (after March 23, 2020), consisting of either in-person, or virtual
* For patients who have had two consecutive video visits, or consecutive telephone visits with supportive care, they will be asked to complete additional questions regarding telehealth visits

Exclusion Criteria:

* Memorial Delirium Assessment Scale (MDAS) of 7 or more or if determined to be of impaired cognition by the clinician at the time of clinic visit as documented in the visit either by history or exam. Providers routinely note screening for mental status with routine administration of the MDAS or history of altered cognition or noted on exam
* Non-English-speaking participants
* Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced cancer seen at the University of Texas MD Anderson Supportive Care Outpatient Clinic
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Assessment of attitudes and beliefs of patients' level of distress and incidence of stressors due to the COVID-19 pandemic, measured by survey. | through study completion, an average of 1 year
  [Survey (COVID Distress Survey) will evaluate overall distress level with degree of increase or decrease assessed on a 7-point Likert scale, with higher scores indicating high distress levels.
Assessment of patients' overall preference and perceptions towards palliative telemedicine vs in person visits during the COVID-19 pandemic. | through study completion, an average of 1 year
  [Survey (Attitudes and beliefs towards telehealth) will evaluate participant preference level with degree of increase or decrease assessed by 5-point Likert scale from "strongly prefer virtual visits" to "strongly prefer in person visits", with high scores indicating preference for in-person visits..

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org